CLINICAL TRIAL: NCT01729702
Title: Evaluation at Rest and Exercise of Clinical, Ultrasonic and Neurohormonal Parameters in Hypertrophic Cardiomyopathies
Brief Title: Neurohormonal Parameters in Hypertrophic Cardiomyopathies
Acronym: REEF-CMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-08
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: 1- Primary (Sarcomeric) Hypertrophic Cardiomyopathy; 2- Obstructive Hypertrophic Cardiomyopathy; 3- Non Obstructive Hypertrophic Cardiomyopathy
Keywords: 1- Hypertrophic cardiomyopathy; 2- BNP; 3- NT-proBNP; 4- Neurohormons
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single group - consecutive patients (Other)
  Interventions: Other: blood sample collection

INTERVENTIONS:
Other: blood sample collection

SUMMARY:
The primary purpose of this study is to demonstrate that changes in plasma levels of circulating neurohormones (mainly BNP and NT-proBNP), measured at rest and post-exercise correlate with exercise functional limitation (assessed by exercise peak VO2) and exercise ultrasonic parameters (as left ventricular filling, obstruction, and mitral regurgitation)

DETAILED DESCRIPTION:
The secondary purposes are to study the kinetics of secretions of natriuretic peptides, and their relationships with extent of MRI myocardial fibrosis with the degree of exercise functional limitation.

ELIGIBILITY:
Inclusion Criteria:

* - Age 18 to 75 years
* Primary (sarcomeric) hypertrophic cardiomyopathy, obstructive or non obstructive, with studies of exercise peak oxygen consumption and cardiac MRI with gadolinium late-enhancement
* Informed consent
* Patient with a social insurance Patient at rest
* - Age 18 to 75 years
* Primary (sarcomeric) hypertrophic cardiomyopathy, obstructive or non obstructive
* Informed consent
* Patient with a social insurance

Exclusion Criteria:

* - Insufficient echogenicity
* Permanent atrial fibrillation
* Complete BBB on the ECG
* LVEF < 35 %
* Previous septal ablation (surgical or percutaneous)
* Simultaneous participation to another biomedical research

If exercise needed:

* contraindication to exercise : hemodynamic instability, uncontrolled high blood pressure (>220/120 mmHg), severe aortic stenosis
* Inability to exercise (muscular, pulmonary, elderly patient)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2009-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Plasmatic Neurohormonal measures: BNP - NT ProBNP - Troponine | Day 1 at rest and during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Albert Hagège, MD-PhD, Study Chair — HEGP - Paris
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France